CLINICAL TRIAL: NCT06768801
Title: Pilot RCT of the Web-app Based Lifestyle Physical Activity Promotion Program (WPAPP) for Middle Aged Latinas
Brief Title: Web-app Based Lifestyle Physical Activity Promotion Program (WPAPP) for Middle Aged Latinas
Acronym: WPAPP-Latina
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Alexandra Garcia, Professor, University of Texas at Austin
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 00007101
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Middle Aged; Women; Depressive Symptoms; Physical Activity; Hispanic or Latino
Keywords: Web-based App
MeSH Terms: conditions — Depression; Motor Activity

STUDY DESIGN:
Intervention Model Description: Two group (intervention and control), random assignment, 3 data collection points
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WPAPP-Latina Intervention (Experimental)
  Interventions: Behavioral: WPAPP-Latina

INTERVENTIONS:
Behavioral: WPAPP-Latina — The WPAPP Latina intervention provides 1) educational information via modules and online resources and 2) coaching via an online forum with a chat function. The educational modules include 11 modules on physical activity promotion and 7 modules on depressive symptoms. The women are also invited to share their experiences with culturally matched interventionists (e.g., Spanish speaking graduate research assistant with expertise in depressive symptoms and physical activity) and with peer participants using a de-identified name in the online chat forum. Participants will be directed to information about physical activity with age-appropriate guidelines from the Centers for Disease Control and Prevention.

SUMMARY:
The purpose of the proposed project is to conduct a pilot randomized controlled trial (RCT) of the Web-App based Lifestyle Physical Activity Promotion Program (WPAPP) for middle-aged Latinas. The WPAPP is a web application (app) to promote lifestyle physical activity that was developed and tested with Korean American middle aged women. It shows promise for effectiveness with Latinas. The specific aims are:

1. To test the feasibility and satisfaction of the WPAPP modified for Latinas.
2. To examine preliminary effectiveness of the WPAPP-Latina on increasing physical activity and decreasing depressive symptoms.

ELIGIBILITY:
Inclusion Criteria: women aged 40-60 who self-identify as Latina or Hispanic women, are able to read and write in English or Spanish, live in the United States, and can use the app and complete online data collection using a smart phone, tablet, or computer.

-

Exclusion Criteria: pregnancy within 3 months of starting the study, having or being of high risk for cardiovascular or musculoskeletal illnesses or injuries

-

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Self-identify as a woman
Enrollment: 40 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Center for Epidemiological Studies - Depression | from baseline to 3 months
  20-item measure of frequency and quantity of depressive symptoms
The modified Barriers to Health Activities Scale | from baseline to 3 months
  16 items scored as 1= never to 4= routinely) about barriers to regular physical activity. Each item asks the women to identify the frequency of interferences with their regular physical activity due to the issue in the individual item. All items will be summed to calculate a total score.
Kaiser Physical Activity Survey | from baseline to 3 months
  Quantity of Physical Activity
Questions on Attitudes Toward Physical Activity, Subjective Norm, Perceived Behavioral Control, and Behavioral Intention | from baseline to 3 months
  The scale is four domains of physical activity; the Attitudes Toward Physical Activity, Subjective Norm, Perceived Behavioral Control, but only the items in the attitude and social influences domains will be used in this study. The attitude domain has six bipolar (-3 to +3) semantic differential scale items. The social influences domain has three unipolar (1 to 7) scale items.
Physical Activity Assessment Inventory | from baseline to 3 months
  13 items measuring self-efficacy related to physical activity in diverse conditions scored from 0= cannot do at all to 100= certainly can do.

IPD SHARING:
Plan to Share IPD: Undecided